CLINICAL TRIAL: NCT00392652
Title: Phase 1 Multiple-Dose Safety, Pharmacokinetic, and Drug Interaction Clinical Study of Nutritional-Grade, Absorption-Enhanced DIM (BR-DIM)
Brief Title: Diindolylmethane in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00867; NCI-2009-00867 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000511393; HSC # 9139; HSC # 9139 (Other: University of Kansas Medical Center); N01-CN-35008-3 (Other: DCP); N01CN35008 (NIH)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy, no Evidence of Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (low-dose oral diindolylmethane) (Experimental): Participants receive low-dose oral diindolylmethane (BR-DIM) twice daily for 4 weeks.
  Interventions: Drug: oral microencapsulated diindolylmethane
- Arm II (high-dose oral diinolylmethane) (Experimental): Participants receive high-dose oral BR-DIM twice daily for 4 weeks.
  Interventions: Drug: oral microencapsulated diindolylmethane

INTERVENTIONS:
Drug: oral microencapsulated diindolylmethane — Given PO
  Other Names: BioResponse DIM; BR-DIM

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of diindolylmethane in healthy volunteers. Chemoprevention is the use of certain drugs or substances to keep cancer from forming, growing, or coming back. The use of diindolylmethane may keep cancer from forming. Collecting and storing samples of blood and urine from healthy volunteers to study in the laboratory may help doctors learn more about the way a person's body handles the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effect of multiple daily dosing with nutritional-grade, absorption-enhanced diindolylmethane (BR-DIM) on the disposition of probe drugs metabolized by cytochrome P4501A2 (CYP1A2) and CYP3A4 in healthy volunteers.

SECONDARY OBJECTIVES:

I. Determine the effect of multiple daily doses of BR-DIM on estrogen metabolites in urine and on activities of CYP2C9, CYP2D6, and P-glycoprotein/OATP.

II. Determine the effect of a single dose of BR-DIM on the disposition of probe drugs that are metabolized or transported by CYP1A2, CYP2C9, CYP2D6, CYP3A4, and P-glycoprotein (P-go).

III. Determine the safety and tolerability of single and multiple daily doses of BR-DIM.

IV. Determine the pharmacokinetics of a single dose of BR-DIM and of the same dose after chronic daily dosing.

V. Determine the pharmacokinetics of a single dose of BR-DIM and of the same dose after chronic daily dosing.

TERTIARY OBJECTIVES:

I. To determine effects of BR-DIM on activities of glutathione-S-transferase (GST), a phase 2 enzyme, in lymphocytes.

OUTLINE: This is a randomized, double-blind study. Participants are stratified according to gender. Participants are randomized to 1 of 2 intervention arms.

Arm I: Participants receive low-dose oral diindolylmethane (BR-DIM) twice daily for 4 weeks.

Arm II: Participants receive high-dose oral BR-DIM twice daily for 4 weeks.

In both arms, participants receive an oral probe-drug cocktail comprising caffeine (CYP1A2), dextromethorphan (CYP2D6), buspirone (CYP3A4), losartan (CYP2C9), and fexofenadine (P-glycoprotein) before randomization and after the first and last dose of BR-DIM.

Blood and urine are collected periodically for pharmacokinetic profiles of BR-DIM and probe drugs.

After completion of study intervention, participants are followed at 1 week.

ELIGIBILITY:
Criteria:

* Healthy men and women
* Nonsmoker confirmed by urine cotinine test
* No active malignancy
* Life expectancy >= 12 months
* Hemoglobin > 10 g/dL
* Absolute granulocyte count > 1,500/mm^3
* Creatinine < 2.0 mg/dL
* Albumin > 3.0 g/dL
* Bilirubin < 1.8 mg/dL
* AST and ALT < 110 U/L
* Alkaline phosphatase < 300 U/L
* Body mass index =< 30
* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective nonhormonal contraception
* No acute, unstable, chronic, or recurring medical conditions
* No strict vegetarians or consumption of > 3 medium servings (1/2 cup each) of cruciferous vegetables per week
* Participants who have stopped eating cruciferous vegetables within the past 2 weeks and agree to refrain from eating them for the duration of the study are eligible
* Cruciferous vegetables include broccoli, cabbage (including coleslaw), cauliflower, bok-choy, brussels sprouts, collards, kale, kohlrabi, mustard greens, rutabaga, turnip, and watercress
* No serious drug allergies or other serious intolerance or allergies
* Mild seasonal allergies allowed
* No chronic conditions, including headaches, dysphoria, fatigue, dizziness, blurred vision, insomnia, rhinorrhea, nausea, vomiting, abdominal pain, diarrhea, constipation, menopausal hot flashes/night sweats, or clinically significant premenstrual syndrome
* No serious acute or chronic illness
* No requirement for chronic drug therapy
* No alcohol ingestion within 48 hours of study treatment
* No investigational drugs within the past 3 months
* No prior chemotherapy
* No concurrent regular medications or hormones
* No recent change in medications or dosage of medications
* No concurrent regular supplements or vitamins
* No concurrent over-the-counter medications
* No concurrent grapefruit or its juice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Effect of diindolylmethane (BR-DIM) on activities of CYP3A4 and CYP1A2 | Up to 1 week
  Descriptive statistics will be calculated on all variables of interest: frequencies and percentages will be used to summarize categorical variables and medians, and ranges will summarize quantitative variables. Paired t-tests will be used to compare enzyme levels post-pre at each dose. Analysis of covariance will be used to determine if there is a dose effect on enzyme levels, using the baseline values as a covariate. If there is no dose effect, the seven subjects at each dose will be pooled which will provide an increase power to detect meaningful changes in enzyme levels.
Grade 2 or higher toxicities, graded using NCI CTC version 2.0 | Up to 1 week
  A one-sided binomial test will be used. Descriptive statistics will be calculated on all variables of interest: frequencies and percentages will be used to summarize categorical variables and medians, and ranges will summarize quantitative variables.
Steady-state pharmacokinetic parameters such as half-life, Cmax, Tmax, and AUC | Up to 1 week
  Pharmacokinetic parameters between pre- and post-menopausal women will be compared using the Wilcoxon rank-sum test.

SECONDARY OUTCOMES:
Drug metabolizing enzyme values (CYP2C9, CYP2D6, P-glycoprotein/OATP, and glutathione-S-transferase) | Up to 1 week
  The probe drug values for the first three enzymes for the baseline (placebo) values and the first-dose BR-DIM values compared to assess inhibitory possible interactions, and between baseline and last-dose BR-DIM values to assess the possibility of either inhibitory or inductive events. Measurements of lymphocyte cytosolic GST activities will compare baseline to last-dose BR-DIM values, and thus assess the possibility of either inhibitory or inductive events. Since we anticipate skewed data, we will compare the values listed above using nonparametric Wilcoxon sign rank tests.
2/16 alpha OHE ratio in urine | Up to 1 month
  A one-way repeated measures analysis of variance will be used to compare this ratio across treatment periods (baseline, one month on BR-DIM, one month after stopping BR-DIM). We will summarize 2/16 alpha OHE ratio at each dose by means and standard deviations. If there is a large degree of skewness the median and range will be utilized as summary measures and Friedman's test utilized to assess the effect of BR-DIM on metabolites of estrogen in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Reed Greg, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States